CLINICAL TRIAL: NCT06951477
Title: Gut Microbiome in Orthopaedics: Investigating the Role of Gut Microbiome Composition in Total Knee Arthroplasty Failure
Brief Title: Gut Microbiome in Orthopaedics: Revision Total Knee Arthroplasty
Acronym: GUMBO
Status: Not yet recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Brent Lanting, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 126857
Record Dates: First submitted 2025-04-07; First posted 2025-04-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Revision Total Knee Arthroplasty; Osteoarthritis, Knee
Keywords: Revision TKA; Gut Microbiome; Implant Loosening; Inflammation; Weight-Bearing Computed Tomography; PET/CT
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect stool samples pre-operatively and at 5 days and 6 weeks post-operatively. Microbial DNA will be extracted from the stool samples and metagenomic sequencing will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Revision TKA: Participants scheduled to undergo a revision TKA will be recruited. They must be more than 3 months post-operation from their primary surgery, and the revision must be for something other than periprosthetic fracture, DAIR (debridement, antibiotics, and implant retention), or stage 2 periprosthetic joint infection.
  Interventions: Procedure: Revision Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Revision Total Knee Arthroplasty — Study participants must be scheduled to receive a revision TKA.

SUMMARY:
Many patients who receive knee replacement surgery must return for a revision (or repeat) surgery due to ongoing pain, stiffness, infection, or implant loosening. The role of the gut microbiome-the collection of bacteria and other microbes within the human gastrointestinal tract-is just beginning to be recognized in orthopaedics. The gut microbiome has been found to affect the immune response and bone regulation, potentially contributing to infection or loosening after total joint replacement. Antibiotics are regularly used in orthopaedic surgery to reduce the risk of infection, yet they might also harm gut microbiota and reduce their potentially beneficial effects. As a result, understanding the relationship between gut microbiota and surgical outcomes has become increasingly important. Therefore, this study aims to determine if there are differences in gut microbiota composition between patients with well-functioning knee replacements and those requiring revision knee replacements. Additional study aims include assessing inflammation, implant loosening, metal ion levels, and circulating bacteria in blood or tissue between well-functioning or failed knee replacements.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a revision TKA
* Willing and able to comply with follow-up requirements
* Ability to provide informed consent
* Ability to read, write, and speak English

Exclusion Criteria:

* Pregnancy
* Less than 3 months post-operation from primary surgery
* Diagnosis of periprosthetic fracture
* Scheduled for DAIR (debridement, antibiotics, and implant retention) revision surgery
* Scheduled for stage 2 PJI revision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at University Hospital scheduled to undergo a revision TKA.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome Composition | Gut microbiome composition will be assessed pre-operatively and at 5 days and 6 weeks post-operation to determine how it changes post-operation.
  The gut microbiome composition of the revision total knee arthroplasty (TKA) cohort prior to revision surgery will be compared to that of the well-functioning TKA cohort. Additionally, we will evaluate changes in the gut microbiome within the revision cohort from before surgery to six weeks after surgery.

SECONDARY OUTCOMES:
Inducible Displacement Measurements with Weight-Bearing Computed Tomography (WBCT) | WBCT exams will be performed at one timepoint prior to the study participant's revision surgery.
  Seated and standing WBCT exams will be performed. The bone and implant will be segmented, and a novel software (WBCT-based radiostereometric analysis (WBCT-RSA)) will be used to measure implant motion between the double seated exams (precision) or seated and standing exams (inducible displacement). Change in implant position will be measured in millimeters as maximum total point motion (MTPM). MTPM will be compared between the revision TKA cohort and a cohort with well-functioning implants.
Inflammation in the Knee Joint Based on [18F]FEPPA Standard Uptake Values (SUV) | PET/CT exams will be performed at one timepoint prior to the study participant's revision surgery.
  Positron Emission Tomography/Computed Tomography (PET/CT) of the knee joint will be performed using the radiotracer [18F]FEPPA, which binds to molecules highly expressed on inflammatory cells. Radiotracer uptake will be quantified using SUV. SUV near the bone and joint will be calculated and compared between the revision TKA cohort and the well-functioning TKA cohort.

OTHER OUTCOMES:
Inducible Displacement and Microbiome Composition | Inducible displacement exams will be performed pre-operatively and will be compared to the gut microbiome from pre-operation to 6 weeks post-operation, and to the intra-operative joint microbiome.
  Joint and gut microbiome composition, along with inducible displacement measurements, will be assessed to determine whether alterations in the gut microbiome lead to increased within-bone implant motion.
Implant Wear Volume and Within-Bone Implant Motion from Inducible Displacement Exams | Inducible displacement exams will be performed pre-operatively and will be compared to the amount of wear that has occurred on implants retrieved during revision surgery.
  Seated and standing WBCT exams will be performed. The bone and implant will be segmented, and a novel software (WBCT-RSA) will be used to measure implant motion between the seated and standing exams (inducible displacement). Change in implant position will be measured in millimeters as MTPM. An optical coordinate measuring machine will be used to quantitatively measure the amount of volume loss from the retrieved implant components. Inducible displacement MTPM will be compared to volume loss to determine if greater within-bone implant motion may cause greater wear of the implant component resulting in more volume loss.
Metal Ion Levels and Within-Bone Implant Motion from Inducible Displacement Exams | Inducible displacement exams will be performed pre-operatively and will be compared to the amount of circulating metal ions pre-operation.
  Seated and standing WBCT exams will be performed. The bone and implant will be segmented, and a novel software (WBCT-RSA) will be used to measure implant motion between the seated and standing exams (inducible displacement). Change in implant position will be measured in millimeters as MTPM. Metal ion levels (cobalt, chromium, nickel, and titanium) will be measured from a blood draw prior to the revision surgery. Inducible displacement MTPM and metal ion levels will be compared to determine if greater within-bone implant motion causes greater levels of circulating metal ions.
[18F]FEPPA Activity and Microbiome Composition | PET/CT exams will be performed pre-operatively and will be compared to the gut microbiome from pre-operation to 6 weeks post-operation, and to the intra-operative joint microbiome.
  Joint and gut microbiome composition will be compared to [18F]FEPPA activity, to assess whether alterations in the gut microbiome contribute to increased inflammation in the knee joint.
[18F]FEPPA Activity and Implant Wear Volume | PET/CT exams will be performed pre-operatively and will be compared to the amount of wear that has occurred on implants retrieved during revision surgery.
  [18F]FEPPA activity from PET/CT will be used to detect the amount of inflammation present in the knee joint. An optical coordinate measuring machine will be used to quantitatively measure the amount of volume loss from the retrieved implant components as an indicator of wear. The relationship between volume loss and [18F]FEPPA activity will be assessed.
[18F]FEPPA Activity and Metal Ion Levels | PET/CT exams will be performed pre-operatively and will be compared to the amount of circulating metal ions pre-operation.
  [18F]FEPPA activity from PET/CT will be used to detect the amount of inflammation present in the knee joint. Metal ion levels (cobalt, chromium, nickel, and titanium) will be measured pre-operatively and the relationship between inflammation and circulating metal ions will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, MD, MSc, FRCSC, Principal Investigator — Schulich School of Medicine & Dentistry
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hext RA, Kaptein BL, Howard JL, Lanting BA, Teeter MG. Inducible displacement of cementless total knee arthroplasty components with conventional and weight-bearing CT-based radiostereometric analysis. J Orthop Res. 2025 Mar;43(3):640-649. doi: 10.1002/jor.26017. Epub 2024 Nov 15. PMID 39545647
- [Background] Xiao PL, Hsu CJ, Ma YG, Liu D, Peng R, Xu XH, Lu HD. Prevalence and treatment rate of osteoporosis in patients undergoing total knee and hip arthroplasty: a systematic review and meta-analysis. Arch Osteoporos. 2022 Jan 14;17(1):16. doi: 10.1007/s11657-021-01055-9. PMID 35029750
- [Background] Li J, Ho WTP, Liu C, Chow SK, Ip M, Yu J, Wong HS, Cheung WH, Sung JJY, Wong RMY. The role of gut microbiota in bone homeostasis. Bone Joint Res. 2021 Jan;10(1):51-59. doi: 10.1302/2046-3758.101.BJR-2020-0273.R1. PMID 33448869
- [Background] Hernandez CJ, Yang X, Ji G, Niu Y, Sethuraman AS, Koressel J, Shirley M, Fields MW, Chyou S, Li TM, Luna M, Callahan RL, Ross FP, Lu TT, Brito IL, Carli AV, Bostrom MPG. Disruption of the Gut Microbiome Increases the Risk of Periprosthetic Joint Infection in Mice. Clin Orthop Relat Res. 2019 Nov;477(11):2588-2598. doi: 10.1097/CORR.0000000000000851. PMID 31283731
- [Background] Chisari E, D'Mello D, Sherman MB, Parvizi J. Inflammatory Bowel Diseases Increase the Risk of Periprosthetic Joint Infection. J Bone Joint Surg Am. 2022 Jan 19;104(2):160-165. doi: 10.2106/JBJS.20.01585. PMID 34648464
- [Background] Hernandez CJ. Musculoskeletal Microbiology: The Microbiome in Orthopaedic Biomechanics. Curr Opin Biomed Eng. 2021 Sep;19:100290. doi: 10.1016/j.cobme.2021.100290. Epub 2021 May 6. PMID 34151053
- [Background] Moran MM, Wessman P, Rolfson O, Bohl DD, Karrholm J, Keshavarzian A, Sumner DR. The risk of revision following total hip arthroplasty in patients with inflammatory bowel disease, a registry based study. PLoS One. 2021 Nov 4;16(11):e0257310. doi: 10.1371/journal.pone.0257310. eCollection 2021. PMID 34735461
- [Background] Abdeen A, Della Valle CJ, Kendoff D, Chen AF. The Paradox of Prosthetic Joint Infection and the Microbiome: Are Some Bacteria Actually Helpful? Arthroplast Today. 2022 Jan 18;13:116-119. doi: 10.1016/j.artd.2021.11.011. eCollection 2022 Feb. PMID 35106346
- [Background] Chisari E, Wouthuyzen-Bakker M, Friedrich AW, Parvizi J. The relation between the gut microbiome and osteoarthritis: A systematic review of literature. PLoS One. 2021 Dec 16;16(12):e0261353. doi: 10.1371/journal.pone.0261353. eCollection 2021. PMID 34914764
- [Background] Hernandez CJ. Musculoskeletal microbiology: The utility of the microbiome in orthopedics. J Orthop Res. 2021 Feb;39(2):251-257. doi: 10.1002/jor.24927. Epub 2020 Dec 7. PMID 33245146
- [Background] Boer CG, Radjabzadeh D, Medina-Gomez C, Garmaeva S, Schiphof D, Arp P, Koet T, Kurilshikov A, Fu J, Ikram MA, Bierma-Zeinstra S, Uitterlinden AG, Kraaij R, Zhernakova A, van Meurs JBJ. Intestinal microbiome composition and its relation to joint pain and inflammation. Nat Commun. 2019 Oct 25;10(1):4881. doi: 10.1038/s41467-019-12873-4. PMID 31653850
- [Background] Moran MM, Wilson BM, Li J, Engen PA, Naqib A, Green SJ, Virdi AS, Plaas A, Forsyth CB, Keshavarzian A, Sumner DR. The gut microbiota may be a novel pathogenic mechanism in loosening of orthopedic implants in rats. FASEB J. 2020 Nov;34(11):14302-14317. doi: 10.1096/fj.202001364R. Epub 2020 Sep 15. PMID 32931052
- [Background] Bourdon CE, Koudys ZJ, Lanting BA, Appleton CT, Thiessen JD, Teeter MG. Attenuation correction for PET/MRI to measure tracer activity surrounding total knee arthroplasty. Eur J Hybrid Imaging. 2022 Nov 7;6(1):31. doi: 10.1186/s41824-022-00152-3. PMID 36336748